CLINICAL TRIAL: NCT00875979
Title: A Phase Ib/II, Open-label Study of the Safety, Tolerability, and Efficacy of Trastuzumab Emtansine (Trastuzumab-MCC-DM1, T-DM1) in Combination With Pertuzumab Administered Intravenously to Patients With Human Epidermal Growth Factor Receptor-2 (HER2)-Positive Locally Advanced or Metastatic Breast Cancer Who Have Previously Received Trastuzumab
Brief Title: A Study of Trastuzumab Emtansine (Trastuzumab-MCC-DM1, T-DM1) in Combination With Pertuzumab Administered to Patients With Human Epidermal Growth Factor Receptor-2 (HER2)-Positive Locally Advanced or Metastatic Breast Cancer Who Have Previously Received Trastuzumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO22495; TDM4373g (Other: Genentech)
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC; Breast Cancer; HER2+; HER2+ breast cancer; HER2 positive breast cancer; herceptin; Trastuzumab emtansine
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; pertuzumab

ARMS (2):
- Trastuzumab emtansine 3.0 mg/kg + pertuzumab 420 mg (Experimental): Patients received trastuzumab emtansine 3.0 mg/kg intravenously (IV) on Day 1 of every 3 week cycle until progressive disease, intolerable toxicity, initiation of another anti-cancer therapy, or patient discontinuation. Patients also received a loading dose of 840 mg of pertuzumab IV on Day 1 of Cycle 1 followed by pertuzumab 420 mg IV on Day 1 of every subsequent 3 week cycle.
  Interventions: Drug: Trastuzumab emtansine [Kadcyla] 3.0 mg/kg; Drug: Pertuzumab 420 mg
- Trastuzumab emtansine 3.6 mg/kg + pertuzumab 420 mg (Experimental): Patients received trastuzumab emtansine 3.6 mg/kg intravenously (IV) on Day 1 of every 3 week cycle until progressive disease, intolerable toxicity, initiation of another anti-cancer therapy, or patient discontinuation. Patients also received a loading dose of 840 mg of pertuzumab IV on Day 1 of Cycle 1 followed by pertuzumab 420 mg IV on Day 1 of every subsequent 3 week cycle.
  Interventions: Drug: Trastuzumab emtansine [Kadcyla] 3.6 mg/kg; Drug: Pertuzumab 420 mg

INTERVENTIONS:
Drug: Trastuzumab emtansine [Kadcyla] 3.0 mg/kg — Trastuzumab emtansine was provided as a single-use lyophilized formulation.
  Other Names: trastuzumab-DM1; trastuzumab-MCC-DM1; T-DM1
  Arms: Trastuzumab emtansine 3.0 mg/kg + pertuzumab 420 mg
Drug: Trastuzumab emtansine [Kadcyla] 3.6 mg/kg — Trastuzumab emtansine was provided as a single-use lyophilized formulation.
  Other Names: trastuzumab-DM1; trastuzumab-MCC-DM1; T-DM1
  Arms: Trastuzumab emtansine 3.6 mg/kg + pertuzumab 420 mg
Drug: Pertuzumab 420 mg — Pertuzumab was provided as a single-use formulation.
  Other Names: Perjeta

SUMMARY:
This was a multi-institutional, multinational, open-label, single-arm Phase Ib/II study designed to evaluate the safety, tolerability, pharmacokinetics, and efficacy of trastuzumab emtansine (trastuzumab-MCC-DM1) administered by intravenous (IV) infusion in combination with pertuzumab in patients with human epidermal growth factor receptor-2 (HER2)-positive locally advanced or metastatic breast cancer who had previously received trastuzumab.

DETAILED DESCRIPTION:
There were 2 phases in the study, a Dose Escalation phase (Phase 1b) and a Dose Expansion phase (Phase 2a). In the Dose Escalation phase, 3 patients were enrolled at the first dose level (3.0 mg/kg trastuzumab emtansine) and and 6 patients were enrolled at the second dose level (3.6 mg/kg trastuzumab emtansine). An additional 58 patients were enrolled at the 3.6 mg/kg trastuzumab emtansine dose level in the Dose Expansion phase (Phase 2a) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented human epidermal growth factor receptor 2 (HER2)-positive locally advanced or metastatic breast cancer.
* Tumor tissue blocks or 15-20 unstained tissue slides for confirmatory central laboratory HER2 status testing and other exploratory assessments.
* Prior trastuzumab in any line of therapy.
* No prior trastuzumab emtansine (T-DM1) or pertuzumab therapy.
* Measurable disease.
* For women of childbearing potential, agreement to use an effective form of contraception and to continue its use for the duration of the study.
* Life expectancy ≥ 90 days.

Exclusion Criteria:

* Less than 21 days since the last anti-tumor therapy, including chemotherapy, biologic, experimental, immune, hormonal, or radiotherapy for the treatment of breast cancer, with the following exceptions: Hormone-replacement therapy or oral contraceptives; palliative radiation therapy involving ≤ 25% of marrow-bearing bone if administered ≥ 14 days prior to first study treatment.
* History of intolerance or hypersensitivity to trastuzumab and/or adverse events related to trastuzumab that resulted in trastuzumab being permanently discontinued.
* Peripheral neuropathy of Grade ≥ 2.
* History of clinically significant cardiac dysfunction.
* Current severe, uncontrolled systemic disease, eg, clinically significant cardiovascular, pulmonary, or metabolic disease.
* Brain metastases that are untreated, progressive, or have required any type of therapy to control symptoms from brain metastases within 60 days of the first study treatment.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine K. Wong, M.Sc., M.D., Study Director — Genentech, Inc.
Locations (19):
- United States (9):
  - Boca Raton, Florida
  - Deerfield Beach, Florida
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Rockville, Maryland
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
- Brussels, Belgium
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec
- France (2):
  - Paris
  - Villejuif
- Cologne, Germany
- Italy (2):
  - Aviano
  - Milan
- Spain (2):
  - Barcelona
  - Valencia

REFERENCES:
- [Derived] Miller KD, Dieras V, Harbeck N, Andre F, Mahtani RL, Gianni L, Albain KS, Crivellari D, Fang L, Michelson G, de Haas SL, Burris HA. Phase IIa trial of trastuzumab emtansine with pertuzumab for patients with human epidermal growth factor receptor 2-positive, locally advanced, or metastatic breast cancer. J Clin Oncol. 2014 May 10;32(14):1437-44. doi: 10.1200/JCO.2013.52.6590. Epub 2014 Apr 14. PMID 24733796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 phases in the study, a Dose Escalation phase (Phase 1b) and a Dose Expansion phase (Phase 2a).
Period: Dose Escalation Phase - 3.0 mg/kg
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient/Legal Guardian Decision | 1 | 0
Period: Dose Escalation Phase - 3.6 mg/kg
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Started | 0 | 6
Completed | 0 | 0
Not Completed | 0 | 6
Not completed — Disease Progression | 0 | 6
Period: Dose Expansion Phase - 3.6 mg/kg
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Started | 0 | 58
Completed | 0 | 11
Not Completed | 0 | 47
Not completed — Disease Progression | 0 | 37
Not completed — Physician Decision | 0 | 3
Not completed — Patient/legal Guardian Decision | 0 | 3
Not completed — Started Non-protocol Anti-Cancer Therapy | 0 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated population: All patients who received at least 1 dose of study drug and had at least 1 follow-up tumor assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg | Total
Number analyzed (Participants) | 3 | 64 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (1.5) | 52.7 (10.8) | 52.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 63 | 66
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: A patient had an objective response if they had a complete response or a partial response on 2 consecutive occasions ≥ 4 weeks apart. For target lesions, a complete response was defined as the disappearance of all target lesions; a partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. For non-target lesions, a complete response was defined as the disappearance of all non-target lesions; a partial response was defined as the persistence of 1 or more non-target lesions.
Time Frame: Baseline through the end of the study (up to 2 years 3 months)
Population: Treated population: All enrolled patients who had baseline measureable disease.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Number analyzed (Participants) | 3 | 64
Percentage of patients | 66.7 [13.5 to 98.3] | 40.6 [28.5 to 53.6]

2. Secondary Outcome: Duration of Objective Response Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Duration of objective response was defined as the time from initial response to disease progression (PD) or death from any cause. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Target lesions should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions.
Time Frame: Baseline through the end of the study (up to 2 years 3 months)
Population: Treated population: All enrolled patients who had baseline measureable disease. Only patients with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Number analyzed (Participants) | 2 | 26
Months | 8.6 [NA to NA] — The confidence interval could not be estimated due to the small sample size. | 13.9 [6.93 to NA] — The upper limit of the confidence interval could not be estimated due to the small sample size.

3. Secondary Outcome: Progression-free Survival Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Progression-free survival was defined as the time from randomization to first documented disease progression (PD) or death due to any cause within 30 days of the last treatment, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Target lesions should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions.
Time Frame: Baseline through the end of the study (up to 2 years 3 months)
Population: Treated population: All enrolled patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Number analyzed (Participants) | 3 | 64
Months | 13.8 [NA to NA] — The confidence interval could not be estimated due to the small sample size. | 6.6 [4.21 to 9.46]

ADVERSE EVENTS:
Time Frame: From informed consent until treatment start (T), serious adverse events (SAE) related to protocol procedures were reported. From the start up to 30 days after the end of T, all AEs and SAEs were reported. Thereafter, only T-related SAEs were reported.
Description: Safety population: All patients who received at least 1 dose of study drug.
Arm/Group | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 22/64
Other Adverse Events (participants affected / at risk) | 3/3 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg (N=3) | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg (N=64)
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Breast cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Osteomyelitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine 3.0 mg/kg + Pertuzumab 420 mg (N=3) | Trastuzumab Emtansine 3.6 mg/kg + Pertuzumab 420 mg (N=64)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 21
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Lacrimation increased (Eye disorders) | 1 | 5
Dry eye (Eye disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 32
Diarrhoea (Gastrointestinal disorders) | 1 | 25
Constipation (Gastrointestinal disorders) | 1 | 21
Vomiting (Gastrointestinal disorders) | 0 | 18
Dyspepsia (Gastrointestinal disorders) | 1 | 11
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 6
Gingival bleeding (Gastrointestinal disorders) | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 3 | 39
Chills (General disorders) | 2 | 20
Pyrexia (General disorders) | 1 | 19
Mucosal inflammation (General disorders) | 0 | 16
Asthenia (General disorders) | 1 | 11
Oedema peripheral (General disorders) | 0 | 7
Chest pain (General disorders) | 0 | 4
Influenza like illness (General disorders) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 5
Sinusitis (Infections and infestations) | 0 | 5
Cellulitis (Infections and infestations) | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 19
Alanine aminotransferase increased (Investigations) | 0 | 18
Blood alkaline phosphatase increased (Investigations) | 0 | 6
Blood bilirubin increased (Investigations) | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Dysgeusia (Nervous system disorders) | 2 | 16
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 16
Headache (Nervous system disorders) | 2 | 16
Dizziness (Nervous system disorders) | 0 | 7
Neuropathy peripheral (Nervous system disorders) | 0 | 7
Insomnia (Psychiatric disorders) | 0 | 15
Depression (Psychiatric disorders) | 1 | 9
Anxiety (Psychiatric disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 5
Hypertension (Vascular disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.